CLINICAL TRIAL: NCT04959266
Title: A Phase I, Open-label, Non-randomised Study to Assess the Effect of Itraconazole (a CYP3A4 Inhibitor), Rifampicin (a CYP3A4 Inducer), and Omeprazole (a Proton Pump Inhibitor) on the Pharmacokinetics of a Single Oral Dose of Adavosertib in Patients With Advanced Solid Tumours
Brief Title: A Study to Assess the Effects of Itraconazole, Rifampicin, and Omeprazole on Pharmacokinetics of Adavosertib
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study terminated because the clinical development programme for Adavosertib has been discontinued
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: D601HC00006
Record Dates: First submitted 2021-06-08; First posted 2021-07-13 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-08

CONDITIONS: Advanced Solid Tumours
Keywords: Proton Pump Inhibitor; Cytochrome P450 3A4 Inhibitor; Cytochrome P450 3A4 Inducer; Pharmacokinetics
MeSH Terms: interventions — adavosertib; Itraconazole; Rifampin; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Patients will receive a single oral dose of adavosertib alone, and a single oral dose of adavosertib concomitantly with itraconazole.
  Interventions: Drug: Adavosertib; Drug: Itraconazole
- Arm B (Experimental): Patients will receive a single oral dose of adavosertib alone, and a single oral dose of adavosertib concomitantly with rifampicin.
  Interventions: Drug: Adavosertib; Drug: Rifampicin
- Arm C (Experimental): Patients will receive a single oral dose of adavosertib alone, and a single oral dose of adavosertib concomitantly with omeprazole.
  Interventions: Drug: Adavosertib; Drug: Omeprazole

INTERVENTIONS:
Drug: Adavosertib — Patients will receive a single dose of Adavosertib orally in arm A, B, and C.
Drug: Itraconazole — Patients will receive Itraconazole orally once daily for 7 days in arm A.
  Arms: Arm A
Drug: Rifampicin — Patients will receive Rifampicin orally once daily for 13 days in arm B.
  Arms: Arm B
Drug: Omeprazole — Patients will receive Omeprazole orally once daily for 5 days in arm C.
  Arms: Arm C

SUMMARY:
This is a Phase 1, open-label, non-randomised, 3-arm (A, B, and C), drug-drug interaction study in patients with advanced solid tumours.

DETAILED DESCRIPTION:
The study will include 3 arms consisting of a screening period of up to 28 days (Day -28 to Day -1), an intervention period (12 days for arm A, 17 days for arm B, and 12 days for arm C), and a follow-up end of treatment [EOT] visit (within 3 days after a 4-day washout period relative to the last dose of adavosertib).

Arm A of this study follows a non-randomised, open-label, 2-intervention design. Patients will receive the following 2 study interventions: a single oral dose of adavosertib alone, and a single oral dose of adavosertib administered concomitantly with itraconazole.

Arm B of this study follows a non-randomised, open-label, 2-intervention design. Patients will receive the following 2 study interventions: a single oral dose of adavosertib alone, and a single oral dose of adavosertib administered concomitantly with rifampicin.

Arm C of this study follows a non-randomised, open-label, 2-intervention design. Patients will receive the following 2 study interventions: a single oral dose of adavosertib alone, and a single oral dose of adavosertib administered concomitantly with omeprazole.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented, locally advanced or metastatic solid tumour, excluding lymphoma, for which standard therapy does not exist or has proven ineffective or intolerable.
2. Eastern Cooperative Oncology Group performance status score of 0 or 1.
3. Predicted life expectancy ≥ 12 weeks.
4. Patients must have normal organ and marrow function at baseline, within 7 days prior to study drug administration.
5. Males and females of childbearing potential who agree to use contraceptive measures must be consistent with clinical study protocol.

Exclusion Criteria:

1. Persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAE] Grade > 2) caused by previous anticancer therapy, excluding alopecia and CTCAE Grade 2 peripheral neuropathy.
2. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of adavosertib, itraconazole, rifampicin, and omeprazole.
3. Any significant cardiac diseases currently or within the last 6 months such as: (a) unstable angina pectoris (b) acute myocardial infarction, congestive heart failure (c) conduction abnormality not controlled with pacemaker or medication (d) significant ventricular or supraventricular arrhythmias.
4. Any of the following:

   1. History or current evidence of congenital long QT syndrome;
   2. concomitant medications known to prolong QT interval or history of medicationrelated QT prolongation.
5. Known to have tested positive for human immunodeficiency virus or active tuberculosis infection.
6. Known active hepatitis infection, positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody, at screening.
7. Any evidence of diseases (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension, renal transplant, active infections, and active bleeding diseases) which prohibit participating in the study.
8. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 4 weeks prior to start of study intervention.
9. Receipt of live virus and live bacterial vaccines whilst the patient is receiving the study intervention and during the 30-day follow-up period. Inactivated flu vaccines are permitted.
10. Use of an anti-cancer treatment drug ≤ 21 days (≤ 6 weeks for nitroureas or mitomycin C) or use of an investigational product within 5 half-lives prior to the first dose of adavosertib.
11. Patient uses drugs that are sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or are moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued 2 weeks or 5 halflives (whichever is longer) prior to Day 1 of dosing.
12. Patients with a known hypersensitivity to adavosertib, itraconazole, rifampicin, and omeprazole or any of the excipients of the product.
13. Currently pregnant (confirmed with positive pregnancy test) or breast-feeding.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Ratios of geometric means of Cmax (maximum observed plasma concentration) when administered in combination with itraconazole/rifampicin/omeprazole relative to adavosertib alone | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of the effect of itraconazole (arm A)/rifampicin (arm B)/omeprazole (arm C) on the Cmax of adavosertib following oral dosing in patients with advanced solid tumours.
Ratios of geometric means of AUCinf (Area under plasma concentration-time curve from time zero to infinity) when administered in combination with itraconazole/rifampicin/omeprazole relative to adavosertib alone | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of the effect of itraconazole (arm A)/rifampicin (arm B)/omeprazole (arm C) on the AUCinf of adavosertib following oral dosing in patients with advanced solid tumours.
Ratios of geometric means of AUClast (Area under the plasma concentration-time curve from zero to time of last quantifiable concentration) when administered in combination with itraconazole/rifampicin/omeprazole relative to adavosertib alone | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of the effect of itraconazole (arm A)/rifampicin (arm B)/omeprazole (arm C) on the AUClast of adavosertib following oral dosing in patients with advanced solid tumours.

SECONDARY OUTCOMES:
Summary of Adavosertib plasma concentrations with time | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of pharmacokinetics (PK) for adavosertib when administered alone and in combination with itraconazole (arm A) /rifampicin (arm B) /omeprazole (arm C).
Descriptive statistics of Cmax | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of Cmax for adavosertib when administered alone and in combination with itraconazole (arm A) /rifampicin (arm B) /omeprazole (arm C).
Descriptive statistics of AUCinf | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of AUCinf for adavosertib when administered alone and in combination with itraconazole (arm A) /rifampicin (arm B) /omeprazole (arm C).
Descriptive statistics of AUClast | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of AUClast for adavosertib when administered alone and in combination with itraconazole (arm A) /rifampicin (arm B) /omeprazole (arm C).
Descriptive statistics of tmax (Time to reach maximum observed concentration following drug administration) | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of tmax for adavosertib when administered alone and in combination with itraconazole (arm A) /rifampicin (arm B) /omeprazole (arm C).
Descriptive statistics of λz (Terminal elimination rate constant) | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of λz for adavosertib when administered alone and in combination with itraconazole (arm A) /rifampicin (arm B) /omeprazole (arm C).
Descriptive statistics of t½λz (Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve) | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of t½λz for adavosertib when administered alone and in combination with itraconazole (arm A) /rifampicin (arm B) /omeprazole (arm C).
Descriptive statistics of CL/F (Apparent total body clearance of drug from plasma after extravascular administration) | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of CL/F for adavosertib when administered alone and in combination with itraconazole (arm A) /rifampicin (arm B) /omeprazole (arm C).
Descriptive statistics of Vss/F (Volume of distribution (apparent) at steady state following extravascular administration) | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of Vss/F for adavosertib when administered alone and in combination with itraconazole (arm A) /rifampicin (arm B) /omeprazole (arm C).
Descriptive statistics of Vz/F (Apparent volume of distribution during the terminal phase after extravascular administration) | Arm A: Days 1-4 and 9-12; Arm B: Days 1-4 and 14-17; Arm C: Days 1-4 and 9-12
  Assessment of Vz/F for adavosertib when administered alone and in combination with itraconazole (arm A) /rifampicin (arm B) /omeprazole (arm C).
Descriptive statistics of Ctrough (Observed lowest drug concentration reached before the next dose is administered) | Arm A: Days 9-11; Arm B: Days 14-17; Arm C: Day 9
  Assessment of Ctrough for itraconazole, rifampicin and omeprazole when administered in combination with adavosertib.
Number of patients with serious and non-serious adverse events | From screening to end of study [within 30 (±7) days of last adavosertib dose]
  Assessment of the safety and tolerability of adavosertib when dosed with itraconazole (arm A), rifampicin (arm B), and omeprazole (arm C).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Research Site, Portland, Oregon
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
- Spain (2):
  - Research Site, Madrid
  - Research Site, Málaga

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the
  Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home